CLINICAL TRIAL: NCT05830162
Title: Oral Antibiotics to Prevent Infection and Wound Dehiscence After Obstetric Perineal Tear - a Double-blinded Placebo Controlled Randomized Trail
Brief Title: Oral Antibiotics After Obstetric Perineal Tear
Acronym: REPAIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hanna Jangö (Other)
Collaborators: Region Hovedstadens Apotek (Other Government)
Responsible Party: Sponsor-Investigator, Hanna Jangö, Prinicipal investigator and sponsor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-501930-49-00
Record Dates: First submitted 2023-03-29; First posted 2023-04-26 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-09

CONDITIONS: Obstetric Trauma; Infections; Wound Dehiscence
Keywords: obstetric tear; women's health; antibiotics; infection; wound dehiscence
MeSH Terms: conditions — Infections | interventions — Amoxicillin; Clavulanic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): The Pharmacy of the main capital region provides the bioclavid (amoxicillin with Clavulanic acid) and placebo tablets for this study. They are responsible for the randomization and packing of the tablets. The randomization will be in randomly variating block sizes.
  Women in the placebo arm will get 3 calcium tablets to take within the fist 24 hours of the delivery. The first tablet must be administrated within 6 hours of the delivery.
  Interventions: Drug: Placebo
- Antibiotics (bioclavid) (Experimental): The Pharmacy of the main capital region provides the bioclavid (amoxicillin with Clavulanic acid) and placebo tablets for this study. They are responsible for the randomization and packing of the tablets. The randomization will be in randomly varying block sizes.
  Women in the antibiotic arm will get 3 tablets bioclavid (amoxicillin and Clavulanic acid) to take within the fist 24 hours of the delivery. The first tablet must be administrated within 6 hours of the delivery.
  Interventions: Drug: Bioclavid (Amoxicillin and Clavulanic acid)

INTERVENTIONS:
Drug: Placebo — We will evaluate how many women gets an infection and/or wound dehiscence after a second degree obstetric tear or episiotomy
  Arms: Placebo
Drug: Bioclavid (Amoxicillin and Clavulanic acid) — We will evaluate how many women gets an infection and/or wound dehiscence after a second degree obstetric tear or episiotomy
  Arms: Antibiotics (bioclavid)

SUMMARY:
The purpose of this study is to investigate if 3 dose of oral antibiotics administrated the first day after a vaginal delivery with a second degree obstetric tear will decrease the risk of infection and/or wound dehiscence compared to women with 3 doses of placebo treatment.

DETAILED DESCRIPTION:
Background:

Obstetric tear occurs in more than 90% of nulliparous women and up to 25% subsequently experience wound dehiscence and/or infection. Some data shows that intravenous antibiotics given during delivery reduces this risk. It is unknown if oral antibiotics given after delivery can reduce the risk of wound dehiscence or infection.

The study-goupe want to investigate whether three doses of antibiotics (amoxicillin 500 mg / clavulanic acid 125 mg) given after delivery can reduce the risk of wound dehiscence and infection.

Methods:

The investigators will perform a randomized, controlled, double-blinded study and plan to include 221 women in each arm with allocation 1:1 in relation to the randomization. The study is carried out at Department of Obstetrics & Gynecology, Herlev University Hospital, Copenhagen, Denmark. The women will be included after delivery if they have had a second-degree tear or episiotomy. The first tabelt has to be taken with in 6 hours from the delivery. After inclusion, the women will have a clinical follow up visit after one week. The tear and healing will be evaluated regarding infection and/or dehiscence. The women will again be invited for a one year clinical examination including ultrasound. Questionaries exploring symptoms related to the vaginal tear and possible complications will be answered at both visits.

The primary outcome is wound dehiscence and/or wound infection, which will be calculated using χ2-tests to compare groups. Secondary outcomes are variables that relate to wound healing, for example pain, use of painkillers, need for further follow-up, as well as other outcomes that may be related to the birth or healing process; urinary or anal incontinence, symptoms of prolapse, female body image and sexual problems.

Discussion:

Reducing the risk of wound dehiscence and/or infection would decrease the number of control visits, prevent the need for longer antibiotic treatment and possibly also decrease both short-term and long-term symptoms. This would be of great importance since the period after a delivery is a crucial time for the whole family.

ELIGIBILITY:
Inclusion Criteria:

* Danish speaking women above 18 years
* Second degree perineal tear and/or episiotomy
* Suturing of obstetric tear at Herlev Hospital

Exclusion Criteria:

* Allergies to the treatment.
* Women who end up with a cesarean-section, including those who have obstetric tears that require stitching or have had an episiotomy
* Women who receive antibiotics intra- or postpartum for other reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Infection in the obstetric tear | Infection will be evaluated 1-2 weeks after the delivery.
  We used the REEDA criteria-Redness, Edema, Ecchymosis, Discharge, and Approximation-to assess this outcome. However, we only diagnosed infection in cases where there was clear clinical evidence, in this study defined as the presence of an abscess or significant wound discharge. In instances of pronounced redness, edema, ecchymosis, or smaller amounts of discharge, these findings were recorded as possible infection or possible resolved infection in the patient's notes as observational comment.
Wound dehiscence | Wound dehiscence will be evaluated 1-2 weeks after the delivery
  We will measure the amount of dehiscence and if above 5 mm it will be diagnoses as a wound dehiscence.

SECONDARY OUTCOMES:
Clinically Relevant Wound Dehiscence | 1-2 weeks post partum
  Throughout the study, we noted a high incidence of wound dehiscence, characterized by a separation of wound edges (diastasis) greater than 5 mm. While some cases were minor, superficial, and without signs of infection, others were more severe. To better assess these more significant cases, we introduced a new secondary outcome: clinically relevant wound dehiscence. This classification was applied to wounds for which the clinician assessed that further follow-up was necessary based on the extent of the dehiscence, the severity of pain, or signs of infection
Pain | 9-12 months after delivery.
  Questionnaire with use of Visual Analogue Scale (VAS) from 1-10 with 10 being the worst pain.
Sexual problems | 9-12 months after delivery.
  Questionnaire
Body image | 9-12 months after delivery.
  Questionnaire -
Number of patients with prolapse | 9-12 months after delivery.
  Gynaecological examination
Prolapse | 9-12 months after delivery.
  Questionnaire (asking if the women have had symptoms of prolapse)
incontinence | 9-12 months after delivery.
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Maternaty ward, Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Perslev K, Klarskov N, Bergholt T, Jango H. Risk of infection and wound dehiscence after use of prophylactic antibiotics in episiotomy or second degree tear (REPAIR study): single centre, double blind, placebo controlled randomised trial. BMJ. 2025 Oct 29;391:e084312. doi: 10.1136/bmj-2025-084312. PMID 41161737
- [Derived] Perslev K, Klarskov N, Bergholt T, Jango H. The REPAIR study: oral antibiotics to prevent infection and wound dehiscence after obstetric perineal tear-a double-blinded placebo controlled randomized trial. Trials. 2024 Mar 27;25(1):221. doi: 10.1186/s13063-024-08069-x. PMID 38532503